CLINICAL TRIAL: NCT06906003
Title: Evaluation of the Impact of Visual Rehabilitation on Anxiety and Depression Severity of Visually Impaired Patients with Advanced Age Related Macular Degeneration
Brief Title: Visual Rehabilitation and Depression in Visually Impaired Patients with AMD
Acronym: RET 06-24
Status: Recruiting | Type: Observational
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Collaborators: Sant'Alessio - Margherita di Savoia (Other)
Responsible Party: Sponsor
Other Study IDs: RET 06-24
Record Dates: First submitted 2025-02-27; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: AMD - Age-Related Macular Degeneration; Anxiety; Depression Disorders
MeSH Terms: conditions — Macular Degeneration; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: visual rehabilitation program — I. meeting: coin recognition II. meeting: reading stories and audio books' listening III. meeting: installation of APPs on their smartphones and tablets and use of voice assistant IV. meeting: management of "table" activities V. meeting: meeting with caregivers.

SUMMARY:
Purpose: The aim of this study is to evaluate the impact of visual rehabilitation in visually impaired patients with advanced AMD by the use of questionnaires on the anxiety and depression status.

Study design: prospective observational study. The study is carried out at the IRCCS Fondazione G.B.Bietti and at the UO Visual Rehabilitation, S. Alessio - Margherita di Savoia.

Study procedures: Visit 1 (screening visit, at IRCCS Fondazione Bietti) After signing the informed consent, all patients received a complete ophthalmological examination, non-invasive diagnostic tests as optical coherence tomography, autofluorescence and microperimetry, and have to complete the questionnaires on the state of anxiety and depression (GAD-7 and PHQ-9).

Visit 2 (at the Sant'Alessio Institute) for a 60-day visual rehabilitation program scheduled in 5 group meetings.

Visit 3 (end-of-study visit, at IRCCS Fondazione G.B. Bietti) complete ophthalmological examination, as per clinical practice, non-invasive diagnostic tests such as microperimetry, optical coherence tomography and autofluorescence and administration of the Patient Health Questionnaire-9 (PHQ-9) questionnaires for depression and the General Anxiety Disorder (GAD-7) questionnaires for anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 55 years
2. Moderate and severe visual impairment (BCVA ≥1/10 and ≤2/10)
3. Diagnosis of advanced non-exudative age-related macular degeneration (AMD)
4. Informed consent freely granted and acquired before the start of the study
5. Ability to understand and willingness to follow the study instructions and procedures

Exclusion Criteria:

1. Visual impairment due to other ocular diseases
2. Mild visual impairment or partial or total blindness
3. Exudative age-related macular degeneration undergoing intravitreal drug treatment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate and severe visually impaired patients affected by non exudative AMD
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Changes of anxiety and depression status in visually impaired patients with AMD undergoing visual rehabilitation program | 12 weeks
  Generalised Anxiety Disorder score (GAD-7, range 0-21,higher scores mean worse outcome) changes after rehabilitation program
Changes of anxiety and depression status in visually impaired patients with AMD undergoing visual rehabilitation program | 12 weeks
  Patient Health Questionnaire score (PHQ-9, range 0-27, higher scores mean worse outcome) changes after rehabilitation program

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione G.B.Bietti, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No